CLINICAL TRIAL: NCT05908721
Title: A Multicenter, Single Arm Phase II Clinical Study Evaluating the Safety of CM310 Recombinant Humanized Monoclonal Antibody Injection in Patients With Seasonal Allergic Rhinitis
Brief Title: Study of CM310 in Patients With Allergic Rhinitis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Keymed Biosciences Co.Ltd (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CM310-107107
Record Dates: First submitted 2023-06-08; First posted 2023-06-18 (Actual); Last update posted 2024-11-08 (Actual); Status verified 2024-06

CONDITIONS: Allergic Rhinitis
MeSH Terms: conditions — Rhinitis, Allergic

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- CM310 (Experimental): Subcutaneous injection
  Interventions: Biological: CM310

INTERVENTIONS:
Biological: CM310 — IL-4Rα monoclonal antibody

SUMMARY:
This study is a multicenter, single arm, open-label phase II clinical study mainly evaluating the safety of CM310 in patients with allergic rhinitis.

DETAILED DESCRIPTION:
Allergic rhinitis (AR) is a non infectious chronic inflammatory disease of the nasal mucosa that is mainly mediated by immunoglobulin E (IgE) in atopic individuals exposed to allergens.

ELIGIBILITY:
Inclusion Criteria:

* Male or female aged 18-65.
* Understand the study and sign the Informed Consent Form voluntarily.
* Take effective contraception measures throughout the study period.

Exclusion Criteria:

* Used other investigational drugs.
* Allergies to drugs with IL-4Rα monoclonal antibody or drug components of CM310.
* Plan to participate in other studies during this clinical trial.
* With malignant or benign tumors of the nasal cavity.
* Other reasons the researcher believes that the subject is not suitable to participate in this study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2023-08-23 (Actual); Primary Completion 2023-12-10 (Actual); Study Completion 2023-12-10 (Actual)

PRIMARY OUTCOMES:
Incidence of adverse events | Week 12
  Incidence (including number of patients, events and percentage) of adverse events.

CONTACTS AND LOCATIONS:
Overall Officials: Luo Zhang, Principal Investigator — Beijing Tong-Ren hospital
Locations (1):
- Beijing Tong-Ren hospital, Beijing, China